CLINICAL TRIAL: NCT01350557
Title: Three Care Models for Elderly Patients With Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Yea-Ing Lotus Shyu, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NHRI-EX98-9404PI; HMRPD180015 (Other: Chang Gung Memorial Hospital)
Record Dates: First submitted 2011-05-06; First posted 2011-05-10 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Hip Fracture
Keywords: Elderly; Hip fracture; Intervention program
MeSH Terms: conditions — Hip Fractures | interventions — Comprehensive Health Care; Subacute Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (No Intervention): Patients receive only usual hospital care
- Subacute care group (Other): Patients receive hospital usual care and subacute care. Subacute care consisted of geriatric consultation, a rehabilitation program, and early discharge planning.
  Interventions: Other: Subacute care
- Comprehensive care group (Experimental): Patients receive not only the subacute care (geriatric consultation, rehabilitation program, and discharge planning), but also health-maintenance interventions to prevent falls, consult on nutrition, and manage depression.
  Interventions: Other: Comprehensive care

INTERVENTIONS:
Other: Comprehensive care — Comprehensive care consisted of subacute care plus health-maintenance interventions to manage depressive symptoms, manage malnutrition, and prevent falls.
  Arms: Comprehensive care group
Other: Subacute care — Subacute care included geriatric consultation, continuous rehabilitation, and discharge planning.
  Arms: Subacute care group

SUMMARY:
Hip fracture in the elderly is associated with excess mortality of 5 to 20%, and mobility problems that usually results in costly hospital stays and lengthy rehabilitation procedures. The purpose of this study is to compare the costs and effectiveness of three care models- acute/sub-acute, comprehensive, and routine care models for hip fractured elders in Taiwan.

DETAILED DESCRIPTION:
Hip fracture in the elderly is associated with excess mortality of 5 to 20%, and mobility problems that usually results in costly hospital stays and lengthy rehabilitation procedures. With this increase in the aging population, hip fracture represents a major and a fast growing health care problem in Taiwan. Currently, the incidence rate of hip fractures is 10 times of the incidence rate for the general population. Despite the use of advanced treatment, the one-year mortality rate (15.4%) remains significant, and many of the patients never recover completely in terms of activities of daily living functions. Many studies in the United States have proved that elderly patients with hip fracture can benefit from post-operative rehabilitation, early discharge planning programs, or transitional care programs. However, little is known about what intervention should be attempted for these patients and their families in Taiwan.

The purpose of this study is to compare the costs and effectiveness of three care models- acute/sub-acute, comprehensive, and routine care models for hip fractured elders in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Admitted to hospital for an accidental single-side hip fracture
* Receiving hip arthroplasty or internal fixation
* Able to perform full range of motion against gravity and against some or full resistance, and have a pre-fracture Chinese Barthel Index (CBI) score >70
* Living in northern Taiwan

Exclusion Criteria:

* Severely cognitively impaired and completely unable to follow orders (determined by a Chinese Mini-Mental State Examination [MMSE] score <10), or
* Terminally ill

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2005-01; Primary Completion 2005-09 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Self-care ability | 1, 3, 6, 12 months after hospital discharge
  Measured by the Chinese Barthel Index (CBI) as ability to perform activities of daily living (ADLs), with scores ranging from 0 to 100.

SECONDARY OUTCOMES:
Depressive symptoms | 1, 3, 6, 12 months after hospital discharge
  Depressive symptoms were assessed using the Chinese version of the Geriatric Depression Scale, short form (GDS-s). Patients with a score ≥ 5 were categorized as at risk for clinical depression.
Nutritional status | 1, 3, 6, 12 months after hospital discharge
  Nutritional status was assessed using the Mini Nutritional Assessment (MNA). MNA scores categorize each person as well-nourished (≥24 points), at risk of malnutrition (17-23.5 points), and malnourished (<17 points).

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Ing L Shyu, PhD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Handoll HH, Cameron ID, Mak JC, Panagoda CE, Finnegan TP. Multidisciplinary rehabilitation for older people with hip fractures. Cochrane Database Syst Rev. 2021 Nov 12;11(11):CD007125. doi: 10.1002/14651858.CD007125.pub3. PMID 34766330
- [Derived] Tseng MY, Liang J, Shyu YI, Wu CC, Cheng HS, Chen CY, Yang SF. Effects of interventions on trajectories of health-related quality of life among older patients with hip fracture: a prospective randomized controlled trial. BMC Musculoskelet Disord. 2016 Mar 3;17:114. doi: 10.1186/s12891-016-0958-2. PMID 26936194
- [Derived] Shyu YI, Liang J, Tseng MY, Li HJ, Wu CC, Cheng HS, Yang CT, Chou SW, Chen CY. Comprehensive care improves health outcomes among elderly Taiwanese patients with hip fracture. J Gerontol A Biol Sci Med Sci. 2013 Feb;68(2):188-97. doi: 10.1093/gerona/gls164. Epub 2012 Sep 7. PMID 22960477